CLINICAL TRIAL: NCT01151293
Title: Personality of Diabetic Patients Will Influence Their Medical compliance-a 5 Years Cohort Follow up With Type D Personality
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Lung Chan, Far-Eastern Memorial Hospital
Other Study IDs: 098011-3
Record Dates: First submitted 2010-06-24; First posted 2010-06-28 (Estimated); Last update posted 2010-06-28 (Estimated); Status verified 2009-07

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type D personality; diabetes; medical compliance; HbA1c; complication; mortality; T2DM
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Diabetes is one of the most common causes of death in Taiwan. With the raising prevalence of diabetes, it became the fourth most common cause of death since 2002. Up to one-tenth of the national health insurance expenditure was used directly in diabetic care. Besides, more expenditure was used in the management of the complications of diabetes, like vascular diseases, renal disease, blindness and neuropathy. Diabetes is a chronic disease, the target treatment is to control HbA1c below 7%, by intensive life style modification, diet control, exercise and medications. Diabetic patient should have a good medical compliance, in order to prevent the tragedy of the complication. A good medical compliance is depended on the individual personality. Personality is the major cause of chronic stress, which is one of the most important cause of psychological stress and the risk factors of the vascular disease and hypertension. Recently, Type D personality had shown the close relationship with patients' prognosis, morbidity, mortality and life quality in different vascular diseases. These vascular diseases are the result of the atherosclerotic process, and diabetes is one of the most important risk factors of the atherosclerotic changes. The investigators believed that type D personality may also affect the medical compliance, the severity (in terms of HbA1c), and the prognosis of diabetic patients. The first part of this study is a cross sectional study, the investigators will try to figure out the relationship of the type D personality toward diabetic medical compliance, and their comorbidity. The second part of this study is a cohort study, base on the population in first part of the study, the investigators will like to construct the correlation of type D personality and diabetic patients' 5-years complication and mortality. The investigators want to establish a more complete vascular care system, improve the medical compliance, lower the complication rates, and improved the quality of life.

ELIGIBILITY:
Inclusion Criteria:

* T2DM patients for OPD
* Age 18-80 y/o
* Inform consent

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: T2DM patients for OPD Age 18-80 y/o Inform consent
Sampling Method: Non-Probability Sample
Dates: Start 2009-07; Primary Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lung Chan, M.D., M. Sc., Principal Investigator — Far Eastern Memorial Hospital